CLINICAL TRIAL: NCT01304732
Title: Totally Implantable Catheters in Pediatric Hematology-oncology: a Study on Infectious Complications
Status: Completed | Type: Observational
Sponsor: Grupo de Apoio ao Adolescente e a Crianca com Cancer (Other)
Responsible Party: Principal Investigator, Orlei Araujo, MD, Grupo de Apoio ao Adolescente e a Crianca com Cancer
Other Study IDs: UTI/IOP 04/11; 0145/11 (Other: CEP UNIFESP)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective analysis of infection on catheters of pediatric oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted between Jan/2008 and Dec/2009

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric oncology patients with diagnosis of catheter infection
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orlei Araujo, MD, Principal Investigator — Grupo de Apoio ao Adolescente e a Crianca com Cancer
Locations (1):
- Grupo de Apoio ao Adolescente e a Criança com Cancer, São Paulo, São Paulo, Brazil